CLINICAL TRIAL: NCT05576753
Title: Prospective Cohort Study on Mesh Shrinkage Measured With MRI After Robot Assisted Laparoscopic Preperitoneal Mesh Repair Using an Iron Oxide Loaded PVDF Mesh
Brief Title: Preperitoneal Umbilical Mesh Area
Acronym: PUMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Maaike Vierstraete, Medical Doctor Department General Surgery, Algemeen Ziekenhuis Maria Middelares
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMA
Record Dates: First submitted 2022-09-25; First posted 2022-10-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Ventral Hernia; Umbilical Hernia; Ventral Incisional Hernia
Keywords: Mesh shrinkage; Abdominal wall surgery
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical | interventions — Herniorrhaphy

STUDY DESIGN:
Intervention Model Description: One single group of 20 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): Patients scheduled for robot assisted laparoscopic preperitoneal repair (vTAPP: ventral transabdominal preperitoneal hernia repair) of a midline ventral hernia
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Procedure: Hernia repair — Robot assisted laparoscopic preperitoneal repair (vTAPP: ventral transabdominal preperitoneal hernia repair) of a midline ventral hernia

SUMMARY:
The aim of this study is to measure the mesh shrinkage and the visualization of the mesh with MRI scan at 1 month and 13 months after robot assisted preperitoneal hernia repair using the visible CICAT mesh (Dynamesh®).

DETAILED DESCRIPTION:
The study will be conducted in the department of surgery in het AZ Maria Middelares, Ghent, Belgium. Dr. Filip Muysoms will personally select and operate all patients eligible for this study. He will inform all patients about the surgery and the follow-up with MRI scan thereafter. Dr. Beckers will perform all MRI examinations of the patients at 1 month and 13 months post-operatively and will be available for questions from the patient.

We want to show that with this type of mesh it is possible to visualize the preperitoneal placed mesh in a safe manner. Furthermore, the positioning of the mesh, mesh shrinkage or mesh shifting will be monitored with this technique. This provides long-term benefit and provides early treatment possibilities in case of post-operative complications related to the mesh position.

ELIGIBILITY:
Inclusion Criteria:

* Primary umbilical hernias up to 2 cm
* Incisional hernias limited to zone M3 (EHS classification) and smaller than 2 cm

Exclusion Criteria:

* <18 years
* Emergency surgery (incarcerated hernia)
* Clean-contaminated, contaminated or dirty procedures (according to the CDC classification)
* Lateral hernias
* Hernias close to the sternum or the pubic bone
* Hernias bigger than 2 cm in diameter.
* Hernias that need a component separation technique.
* Previous mesh repair on the midline
* ASA score> 4
* Pregnancy
* No patient Informed Consent
* Life expectancy of less than 2years
* Contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of mesh surface (percentage) | 1 month and 13 month post-operatively
  Shrinkage rate / change of the mesh surface (percentage) as measured with the MRI between 1 month and 13 months postoperatively, defined as (100 - mesh surface at 13 months x 100 / mesh surface at 1 month)

SECONDARY OUTCOMES:
Change in mesh surface between implantation surface size | 1 month and 13 month post-operatively
  Change in mesh surface between implantation surface size, surface at 1m and at 13m
Change in mesh width and length between implantation surface size | 1 month and 13 month post-operatively
  Change in mesh width and length between implantation surface size, surface at 1m and at 13m
Operation duration | once during operation
  Recording of the operation duration needed for robot-assisted ventral TAPP procedure
Intra-operative complications | until 4 weeks post-operative
  Intra-operative complications registered until 4 weeks after the hernia repair
Early post-operative complications | until 30 days post-operative
  Early post-operative complications detected until 30 days after hernia repair
Late complications | After 30 days post-operative
  Late complications (after 30 days)
Quality of Life questionnaire | Preoperatively, 30 days, 13 months
  Minimum score is 0, maximum score is 90. The higher the score, the worse the outcome
Body image score | Preoperatively, 30 days, 13 months
  Minimum score is 0, maximum score is 10. A higher score means a higher level of body image disturbance (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Maaike Vierstraete, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium